CLINICAL TRIAL: NCT06860009
Title: Psychological Intervention for Fatigue in Inflammatory Bowel Diseases: a Randomized Controlled Trial
Brief Title: Psychological Intervention for Fatigue in Inflammatory Bowel Diseases
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PEARL
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: IBD; Crohn's Diseases; Ulcerative Colitis (UC)
Keywords: fatigue; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Fatigue | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in early or late intervention group. The early intervention group immediately start with the intervention, while the late intervention group will wait until week 28 to start with the 14 week intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention group (Other): Group starts immediately with the 14-week intervention
  Interventions: Behavioral: Multicomponent psychological intervention; Behavioral: Early start
- Late intervention group (Other): Group starts with 14-week intervention after 28 weeks
  Interventions: Behavioral: Multicomponent psychological intervention; Behavioral: Late start (after 28 weeks)

INTERVENTIONS:
Behavioral: Multicomponent psychological intervention — The multicomponent intervention starts with 8 sessions of ACT (Acceptance and commitment therapy) once a week. After four weeks, patients start with graded activity and frequent napping. After eight weeks in the intervention period, patients will have consults with an IBD psychologist every two weeks. The intervention period is 14 weeks in total.
Behavioral: Early start — Patients in the early group immediately start with the multicomponent psychological intervention
  Arms: Early intervention group
Behavioral: Late start (after 28 weeks) — Patients in the late intervention group will wait 28 weeks before starting the intervention
  Arms: Late intervention group

SUMMARY:
The investigators would like to evaluate the effect of a multicomponent psychological treatment on fatigue as a symptom of patients with inflammatory bowel diseases (IBD). The intervention will be a combined program consisting of a psychological intervention (Acceptance and Commitment Therapy) and a behavioral intervention (implementation of frequent short naps and graded increase of physical activity). Next to the hypothesized effect on fatigue, the investigators will also measure the effect on fatigability, IBD related disability, anxiety, depression, stress, disease acceptance and perceived control as well as (biomarkers of) disease activity.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) and Crohn's disease (CD) are chronic inflammatory bowel diseases that significantly impact patients' quality of life. One of the most prevalent and distressing symptoms associated with both UC and CD is fatigue, which can arise from both the physiological effects of the diseases and the psychological burden of living with a chronic condition. Despite the importance of addressing fatigue, traditional treatment approaches often focus primarily on physical symptoms, neglecting the multifaceted nature of fatigue that includes emotional and lifestyle factors.

This research aims to evaluate a novel multicomponent intervention that combines Acceptance and Commitment Therapy (ACT), frequent napping, and Graded Activity. Each component targets different dimensions of fatigue:

Acceptance and Commitment Therapy (ACT): ACT is a mindfulness-based therapeutic approach that encourages individuals to accept their thoughts and feelings rather than fighting against them. It promotes psychological flexibility and helps individuals commit to actions aligned with their values, even in the presence of discomfort. Previous studies have demonstrated ACT's effectiveness in managing chronic pain, anxiety, and other health-related issues, suggesting its potential benefit in addressing fatigue in chronic conditions like UC and CD.

Frequent Napping: Napping has been shown to help mitigate daytime fatigue, improve alertness, and enhance overall well-being. For patients with UC and CD, who often experience irregular sleep patterns due to their symptoms, implementing structured napping could serve as a valuable strategy for managing fatigue. However, this may be less suitable for patients working fulltime.

Graded Activity: Graded Activity is a structured approach to increase physical activity gradually. It involves setting achievable goals and progressively increasing activity levels, which can help mitigate fatigue and improve overall physical functioning. In the context of UC and CD, where patients may experience cycles of flare-ups and remission, Graded Activity can provide a tailored strategy to reintroduce physical activity safely and effectively.

The rationale for combining these three interventions lies in their complementary nature. While ACT addresses the psychological and emotional aspects of fatigue, frequent napping provides immediate relief and recovery opportunities. Graded Activity contributes a structured method for increasing physical activity, helping patients regain their strength and stamina over time. Together, these components create a comprehensive framework that addresses fatigue from multiple angles, which is essential given the complex interplay of physical, emotional, and behavioral factors in both UC and CD.

This research has the potential to make significant contributions to the management of fatigue in patients with UC and CD. By integrating psychological, physiological, and behavioral strategies, the multicomponent intervention could offer a holistic approach that enhances patient care. The findings could inform clinical practice, paving the way for more tailored, multidisciplinary interventions that address the diverse needs of individuals with chronic illnesses.

In conclusion, this study seeks to bridge the gap in existing research by exploring the combined effects of ACT, frequent napping, and Graded Activity on fatigue in patients with UC and CD. The results could lead to improved therapeutic strategies, ultimately enhancing the quality of life and well-being of those living with these challenging conditions.

Patient (eligibility criteria) Inclusion criteria are being at least 18 years and younger than 70 years of age, a diagnosis of CD, UC or IBD type unclassified (IBDU), more than one year of follow-up since diagnosis, no new IBD medication (mesalamine, steroids, thiopurines, methotrexate, biologicals or small molecules) in the past three months prior to baseline, no objective signs of active disease (CRP <10 mg/L AND faecal calprotectin <250 µg/g), a score of <30 on the FACIT Fatigue scale, no planned surgery during the study, no iron (<65 µg/dL), vitamin D (<11 µg/L) , vitamin B12 (<197 ng/L) or folic acid (<3.9 µg/L) deficiency or malnutrition (weight loss >10-15% within six months, BMI <18.5 kg/m², NRS >5 and serum albumin <30 g/L) , no BMI >30 kg/m², no thyroid dysfunction, no hypophosphatemia (<0.64 mmol/L), no physical injury (according to researcher's interpretation), no self-reported sleep disturbance or apnea diagnosis, no present or past severe psychiatric disease diagnosis (ongoing major depression, schizophrenia, bipolar disease, ongoing substance abuse), no new psychotropic medication or change of dosage in the past three months prior to baseline, possessing a smartphone, availability to commit to daily behavioral changes, and being fluent in Dutch. Furthermore, patients will be asked to sign an informed consent.

Intervention The intervention is a combined program incorporating ACT alongside a behavioral approach that emphasizes frequent napping and a gradual increase in physical activity.

ACT is a psychological approach focused on accepting aspects beyond personal control while committing to actions that enhance and enrich one's life. This therapy utilizes strategies of acceptance and mindfulness, combined with commitment and behavior change techniques, to foster psychological flexibility. Key processes in ACT include acceptance, cognitive defusion, committed action, present-moment awareness, self-as-context, and values. The program will be specifically tailored to address fatigue related to IBD and will consist of eight weekly one-hour individual sessions.

1. Introduction to ACT: Overview of ACT principles, emphasizing mindfulness and acceptance in the context of IBD fatigue.
2. Understanding Fatigue: Exploration of the individual's experience with fatigue, including its impact on daily life and emotional well-being.
3. Mindfulness Skills: Teaching mindfulness techniques to help individuals stay present and manage fatigue-related thoughts and feelings.
4. Values Clarification: Identifying personal values and goals to enhance motivation and provide direction despite fatigue.
5. Acceptance Techniques: Learning to accept the reality of fatigue rather than struggling against it, fostering a compassionate attitude toward oneself.
6. Cognitive Defusion: Strategies to create distance from unhelpful thoughts related to fatigue, reducing their impact.
7. Behavioral Activation: Developing a plan for gradually engaging in valued activities, tailored to energy levels and limitations.
8. Review and Future Planning: Reflecting on progress, reinforcing skills learned, and creating a long-term strategy for managing fatigue and maintaining well-being.

After four weeks, participants will begin a personalized exercise regimen that includes frequent naps and gradually increasing activity levels. Participants will be encouraged to take two to five naps (depending on fatigue severity), each lasting 15 to 20 minutes, interspersed with active periods. "Active" refers to any non-resting or non-sleeping activity, which means that reading or watching TV is also considered active. Provided the participant reports an increase in energy, the amount of naps can be tapered off, while nap durations always remain consistent.

To establish a baseline for the graded activity program, participants will record their walking (or cycling, based on their preference) over five days (not necessarily consecutive), noting the duration each day until significant pain, fatigue, or shortness of breath occurs. This will help determine the maximum time at five different points. The average of these measurements will inform the initial activity level. In the first week of the intervention, participants will engage in walking three times at 80% of the average time achieved. Afterward, activity time will increase by 10-15% weekly. For those accustomed to regular exercise, running may replace walking or cycling, following the same protocol.

The overall intervention will span 14 weeks. Following the eight ACT sessions, participants will have two-weekly individual follow-up consultations with an IBD psychologist for ongoing support regarding napping and graded activity.

For data collection, participants will wear a smartwatch to track their activity levels. This data will serve solely as a measurement tool for researchers, and participants will not have access to their own activity data.

Comparison This study will be a prospective, randomized-controlled, monocentric, superiority trial utilizing a waiting list with a treatment-as-usual control arm. Half of the participants will start with the psychological intervention immediately (early intervention group), while the other half will wait six months before starting the intervention (late intervention or control group).

Outcome The primary endpoint is the percentage of participants achieving a ≥20% improvement on the FACIT Fatigue Scale (indicating reduced fatigue) between baseline and week 14. The FACIT Fatigue Scale is a brief 13-item tool that evaluates fatigue experienced during daily activities over the past week. Fatigue is rated on a four-point Likert scale (4 = not at all fatigued to 0 = very fatigued). Total scores range from 0 to 52, with lower scores indicating higher fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Males and females 18-70 years old.
3. Patients with a diagnosis of ulcerative colitis (UC), Crohn's disease (CD), inflammatory bowel disease type unclassified (IBDU) based on radiology, endoscopy and/or histology
4. Patients with a disease duration of more than one year
5. Patients with a score of <30 on the FACIT Fatigue scale
6. Patients possessing a smartphone
7. Patients with an availability to commit to daily behavioural changes
8. Patients being fluent in Dutch.

Exclusion Criteria:

1. Patients that initiated new IBD medication (steroids, mesalamine, thiopurines, methotrexate, biologicals or small molecules) in the past three months prior to screening
2. Patients with objective signs of active disease (CRP<10mg/L or faecal calprotectin <250µg/g) at screening
3. Participation in an interventional Study with an investigational medicinal product (IMP) or device at screening
4. Patients with planned surgery at screening
5. Patients with an iron (<65 µg/dL), vitamin D (<11 µg/L), vitamin B12 (<197 ng/L) or folic acid (<3.9 µg/L) deficiency or malnutrition (weight loss >10-15% within six months, BMI <18.5 kg/m², NRS >5 or serum albumin <30 g/L) at screening
6. Patients with thyroid dysfunction or hypophosphatemia at screening
7. Patients with physical injury (according to researcher's interpretation) at screening
8. Patients with self-reported sleep disturbance or periods of apnoea at screening
9. Patients with BMI >30 kg/m² at screening
10. Patients with present or past diagnosis of severe psychiatric disease diagnosis (ongoing major depression, schizophrenia, bipolar disease, ongoing substance abuse) at screening
11. Patients that initiated new psychotropic medication or had a changed dosage of psychotropic medication in the past three months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
FACIT fatigue scale | 14 weeks
  The percentage of participants achieving a ≥20% improvement on the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (indicating reduced fatigue) between baseline and week 14.